CLINICAL TRIAL: NCT05753995
Title: Imaging of Proinflammatory Activated Microglia Using Purine 2X7 (P2X7) Receptor Scintigraphy in Immuno-Positron Emission Tomography (PET) Scanner in Glioblastoma Patients: a Proof-of-principle Imaging Study
Brief Title: Immuno-Positron Emission Tomography (PET)-Glioma Study, a Proof-of-principle Imaging Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Immuno-PET-Glioma study
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other): for diagnostic
  Interventions: Diagnostic Test: PET imaging

INTERVENTIONS:
Diagnostic Test: PET imaging — The evaluation of PET imaging using PET ligand [18F]JNJ-64413739 or a [18F] labeled equivalent in vivo in patients.

SUMMARY:
Imaging of proinflammatory activated microglia by Purine 2X7 (P2X7) receptor scintigraphy in Positron Emission Tomography (PET) scanner in Glioblastoma patients.

DETAILED DESCRIPTION:
Glioblastomas are extremely malignant tumors of the brain; despite different therapeutic approaches, the median survival is only about 1 ½ years. This makes the need for action to investigate the mechanisms of action of new drug approaches all the more urgent. In the therapy of malignant intracerebral neoplasms, immunological processes between tumor and endogenous immune response represent a key phenomenon for understanding response.

In the CheckMate-143 trial, an anti-programmed cell death-1 monoclonal antibody disappointed by ineffectiveness in the vast majority of Glioblastoma patients (although a minority benefited significantly). This will be largely explained by the immunological milieu of the tumor. One-third of the cells in Glioblastoma constitute the microglia or monocyte cell population. These immunocompetent cells also serve as a protective shield for the Glioblastoma against a possible therapy-induced endogenous immune response.

Corresponding research is being conducted preclinically on cell cultures, brain tissue samples (immunohistochemistry, autoradiography) and in animal models. A major role is played by microglial cells, which perform the immunocompetent function in the brain. Microglia and monocytes have an activation state as well as an opposite of a suppressive one in their immunological function. This M1 or M2 concept is similar to the old postulated Th1 or Th2 principle in lymphocytes. Different purinergic receptors -P2Y12R and Purine receptor 2XR - are active here, respectively. Recently, antibody-based positron-emitter-labeled tracers have been developed for this purpose and thus, in principle, positron emission tomography (PET) imaging in vivo is possible.

The subsequent clinical relevance of a better understanding of these processes would consist in a combined therapeutic concept, in which additionally an immunomodulation in the desired direction of the regional activity of the immunocompetent cells could take place.

Methods for in vivo imaging of activated microglia in positron emission computed tomography scanners (PET) have already been developed - e.g. translocator protein positron emission tomography (TSPO-PET) by detecting mitochondrial activation of microglial cells. Here, however, it is not possible to distinguish between pro- and anti-inflammatory function of the immunocompetent cells. However, it is possible to do so by specific receptor recognition. For example, the purinergic receptor P2X7 is only expressed during proinflammatory activity. For this purpose, the positron emission tomography scanners (PET) tracer [18-Fluorine] Johnson & Johnson (JNJ)-64413739 has been developed in the academic research field. Patient cohort studies are still pending in this regard. Our intention is to investigate in patients with untreated Glioblastoma whether effective imaging of immunological disease activity is possible in this way.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new probable diagnosis of glioblastoma based on MRI imaging.
* prior to initiation of specific tumor therapy and prior to any surgery (including biopsy)
* short-term medication for cerebral edema (including corticosteroids) and short-term administration of antiepileptic drugs are not a reason for exclusion

Exclusion Criteria:

* Non-business capacity
* Pregnancy
* breastfeeding period
* Other malignant disease (active)
* Concurrent participation in another clinical trial
* Foreseeable compliance problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Immuno PET can be used to visualize the immunological environment of the tumor (Glioblastoma). | 1-2 years
  Thus, the aim of the pilot study, which follows an exploratory approach, is to evaluate PET imaging in vivo in patients using PET ligand [18F]JNJ-64413739 or a [18F] labeled equivalent.
  To evaluate if it is possible to visualize (visually topically deniable increased Tracer-uptake) the immunological processes in tumor or adjacent brain structures in sufficient image quality.
  We practice measurement by SUV (= standard uptake value) of the morphologically identified glioblastoma lesion relative to normal brain tissue: TBR (=tumor background ratio) - as a quantification of immunological processes inside the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pichler, PD, MD, Principal Investigator — Kepler University Hospital
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria